CLINICAL TRIAL: NCT07326371
Title: A Single-Center, Prospective Study Evaluating the Efficacy and Safety of Glofitamab Combined With CAR-T Therapy in Patients With High-Risk Relapsed/Refractory Large B-Cell Lymphoma
Brief Title: Glofitamab Combined With CAR-T Therapy in R/R DLBCL
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Glofit_peri_CART
Record Dates: First submitted 2025-12-26; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-07

CONDITIONS: DLBCL - Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Dendritic Cell Sarcoma, Interdigitating | interventions — glofitamab; obinutuzumab; axicabtagene ciloleucel; relmacabtagene autoleucel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Glofit_CART (Experimental): After undergoing leukapheresis, patients will receive treatment in three phases: the bridging phase, the CAR-T treatment phase, and the consolidation phase.
  Bridging Phase:
  All patients will receive two cycles of Glofitamab treatment. On Day 1 of Cycle 1, patients will receive 1000 mg of Obinutuzumab as pretreatment.
  After the completion of Cycle 2, patients will undergo an assessment.
  CAR-T Treatment Phase:
  Participants will receive lymphodepletion therapy with the FLU/CY regimen from Day -5 to Day -3.
  On Day 0, patients will receive the CAR-T cell infusion.
  Consolidation Phase:
  Based on the efficacy assessment on Day 28, the subsequent treatment plan will be determined: Patients achieving complete response (CR) will not receive additional Glofitamab treatment.
  Patients with partial response (PR), stable disease (SD), or progressive disease (PD) will continue to receive Glofitamab treatment for four additional cycles.
  Interventions: Drug: Glofitamab; Drug: Obinutuzumab; Drug: Axicabtagene Ciloleucel; Drug: Relmacabtagene autoleucel (relma-cel)

INTERVENTIONS:
Drug: Glofitamab — Glofitamab IV infusion will be administered as per the schedule specified in the respective arm.
Drug: Obinutuzumab — Obinutuzumab IV infusion will be administered as per the schedule specified in the respective arm.
Drug: Axicabtagene Ciloleucel — Axicabtagene Ciloleucel IV infusion will be administered as per the schedule specified in the respective arm.
Drug: Relmacabtagene autoleucel (relma-cel) — Relmacabtagene autoleucel IV infusion will be administered as per the schedule specified in the respective arm.

SUMMARY:
This study is a single-center, open-label, prospective study aimed at evaluating the efficacy and safety of Glofitamab combined with CAR-T therapy in patients with high-risk relapsed/refractory large B-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Histologically confirmed large B==cell lymphoma with CD19 and CD20 expression, including diffuse large B==cell lymphoma (DLBCL) not otherwise specified (NOS); primary mediastinal large B==cell lymphoma (PMBCL); high==grade B==cell lymphoma (HGBL); and DLBCL transformed from follicular lymphoma
* Patients who have relapsed after at least one prior line of therapy or are refractory, including those who have received anthracycline==containing chemotherapy regimens and anti==CD20 monoclonal antibody therapy
* Patients must be willing to receive CAR==T and Glofitamab therapy and be deemed suitable for CAR==T and Glofitamab treatment by the investigator
* Presence of at least one high==risk prognostic factor: (1) extranodal involvement; (2) maximum tumor diameter > 4 cm; (3) TP53 mutation
* No CNS involvement
* ECOG Performance Status of 0, 1, or 2
* Life expectancy ≥12 weeks
* Adequate hematologic function (unless due to underlying disease, such as extensive bone marrow involvement, or secondary to lymphoma==related splenomegaly as determined by the investigator, but transfusion of blood products is allowed) and adequate liver, renal, pulmonary, and cardiac function, defined as follows:

  * Neutrophil count ≥ 1.0 × 10^9/L, platelet count ≥ 50 × 10^9/L, lymphocyte count ≥ 0.1 × 10^9/L
  * ALT/AST ≤ 2.5 × ULN and total bilirubin < 1.5 × ULN (except for participants with Gilbert's syndrome or lymphoma involvement of the liver)
  * Creatinine clearance ≥ 30 mL/min
  * Pulmonary function: ≤ CTCAE grade 1 dyspnea, oxygen saturation (SpO2) ≥ 92% on room air
  * Cardiac function: LVEF ≥ 40%
* Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to initiating study treatment. Women who are postmenopausal (defined as no menses for ≥ 12 months without an alternative medical cause) or have undergone surgical sterilization (removal of ovaries and/or uterus) are not required to undergo a pregnancy test
* For female participants of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception, and agree to refrain from donating eggs
* For male participants: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods, and agree to refrain from donating sperm
* Patients with a distant history of autoimmune disease or well==controlled autoimmune disease may be eligible for enrollment at the investigator's discretion

  * Patients with a history of autoimmune==related hypothyroidism who are on a stable dose of thyroid replacement hormone may be eligible for this study
  * Patients with a history of disease==related immune thrombocytopenic purpura or autoimmune hemolytic anemia may be eligible for this study
  * Patients with a history of type 1 diabetes mellitus who are well controlled (defined as hemoglobin A1c < 8% at screening and no episodes of diabetic ketoacidosis) are eligible for this study
  * Patients with eczema, psoriasis, chronic lichen simplex, or vitiligo with only skin involvement (e.g., excluding psoriatic arthritis) are eligible for this study if they meet all of the following conditions： Rash must cover < 10% of body surface area The disease is well controlled at baseline and only requires low==potency topical corticosteroids No acute exacerbations of an underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologics, oral calcineurin inhibitors, or high==potency oral corticosteroids within the past 12 months
* Subjects with a history of stroke who have not experienced a stroke or transient ischemic attack in the past 2 years and have no residual neurological deficits, as determined by the investigator, may participate in this study

Exclusion Criteria:

* History of allergic reactions to compounds with similar chemical or biological composition to axi==cel, relma==cel, glofitamab, obinutuzumab, or other drugs used in the study.
* Active or uncontrolled infections requiring systemic therapy (including fungal, bacterial, viral, etc.)
* History of allogeneic hematopoietic stem cell transplantation
* History of organ transplantation
* Viral infections deemed uncontrollable by antiviral medications, as determined by the investigator, including:

  * Active hepatitis B virus (HBV) infection with HBV DNA ≥ 500 IU/mL (2500 copies/mL)
  * Positive hepatitis C virus (HCV) RNA test
  * Positive human immunodeficiency virus antibody (HIV==Ab) test
  * Positive Treponema pallidum antibody (TP==Ab) test
  * Cytomegalovirus (CMV) DNA levels above the upper limit of normal
  * Epstein==Barr virus (EBV) DNA levels above the upper limit of normal
* Current or past history of CNS disease, such as stroke, epilepsy, CNS vasculitis, or neurodegenerative disease
* Presence of brain metastases or active primary central nervous system lymphoma
* Significant or extensive history of cardiovascular disease such as New York Heart Association Class III or IV cardiac disease or Objective Assessment Class C or D, myocardial infarction within the last 6 months prior to the start of Cycle 1, unstable arrhythmias, or unstable angina
* Presence of severe genetic disorders or severe autoimmune diseases, including but not limited to myocarditis, pneumonitis, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid syndrome==associated vascular thrombosis, Wegener's granulomatosis, Sjögren's syndrome, Guillain==Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis
* Known or suspected history of hemophagocytic lymphohistiocytosis (HLH)
* Thromboembolic events (e.g., myocardial infarction, pulmonary embolism, deep vein thrombosis, or other systemic embolic events) within 6 months prior to screening
* Malignancies other than the indication for this trial within 5 years prior to screening, except for in situ cancers (e.g., cervical, bladder, breast) or non==melanoma skin cancers
* Receipt of chemotherapy drugs, tumor radiotherapy, or immunosuppressive antibodies such as anti==TNF, anti==IL6, or anti==IL6R within 4 weeks or 5 half==lives (whichever is shorter) prior to mononuclear cell collection
* Vaccination with live, attenuated vaccines within 3 months prior to mononuclear cell collection, or expected need for such vaccination during the trial
* Currently pregnant or breastfeeding, or planning to become pregnant during the study or within 12 months after the last dose
* Patients currently participating in other clinical trials (e.g., new drug clinical trials, registration studies, investigator==initiated clinical studies)
* Deemed unsuitable for this clinical trial by the investigator (e.g., poor compliance, substance abuse)
* Evidence of significant, uncontrolled concomitant diseases that could affect compliance with the study protocol or interpretation of results
* Any other diseases, metabolic dysfunctions, physical examination findings, or clinical laboratory results that reasonably suggest the presence of a condition that contraindicates the use of the investigational drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Complete Response Rate (CRR) | Baseline up to the end of treatment (EOT) (approximately 4 months)
  Assessed by Investigator per Lugano Response Criteria for Malignant Lymphoma

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Baseline up to the EOT (approximately 4 months)
  Assessed by Investigator per Lugano Response Criteria for Malignant Lymphoma
Duration of Response (DoR) | From the date of the first occurrence of a documented CR or partial response (PR) to the date of progression, relapse, or death from any cause, whichever occurs first (up to approximately 42 months)
PFS | From the start of treatment until the first occurrence of disease progression or relapse, or death from any cause, whichever occurs earlier (approximately 42 months)
  Assessed by Investigator per Lugano Response Criteria for Malignant Lymphoma
Overall Survival (OS) | From the start of treatment until the date of death from any cause (approximately 42 months)
Number of Participants with TEAEs | Up to the end of the study (approximately 42 months)
  Incidence and severity of adverse events, with severity determined according to the NCI CTCAE v5.0 grading scale, including CRS, with severity determined according to the ASTCT CRS grading criteria